CLINICAL TRIAL: NCT06519266
Title: A Phase III Randomized Controlled Multicentre Trial of Percutaneous Hepatic Perfusion in Combination With Ipilimumab and Nivolumab Compared to Ipilimumab and Nivolumab Only in Patients With Uveal Melanoma Liver Metastases
Brief Title: PHP in Combination With IPI1/NIVO3 Compared to IPI3/NIVO1 Only in Patients With Uveal Melanoma Liver Metastases
Acronym: SCANDIUM-III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508156-20-00
Record Dates: First submitted 2024-07-10; First posted 2024-07-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Uveal Melanoma; Liver Metastases
Keywords: Percutaneous Hepatic Perfusion; Immunotherapy; Uveal Melanoma; Liver metastases; SCANDIUM III trial
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IPI3/NIVO1 (Active Comparator): Patients will be treated with 4 cycles of intravenous (i.v.) infusion with ipilimumab 3mg/kg and nivolumab 1mg/kg q3w followed by continued i.v. nivolumab 480mg q4w up to 1 year
  Interventions: Drug: IPI3/NIVO1
- PHP + IPI1/NIVO3 (Experimental): Patients will be treated with two cycles of PHP (CHEMOSAT® Hepatic Delivery System for Melphalan) six weeks apart, followed by two cycles of i.v. ipilimumab 1mg/kg and nivolumab 3mg/kg q3w, followed by continued i.v. nivolumab 480mg q4w up to 1 year
  Interventions: Device: PHP; Drug: IPI1/NIVO3

INTERVENTIONS:
Device: PHP — Patients will be treated with 2 cycles of PHP (CHEMOSAT® Hepatic Delivery System for Melphalan) six weeks apart
  Other Names: CHEMOSAT® Hepatic Delivery System for Melphalan
  Arms: PHP + IPI1/NIVO3
Drug: IPI1/NIVO3 — Patients will be treated with 2 cycles of i.v. ipilimumab 1mg/kg and nivolumab 3mg/kg q3w, followed by continued i.v. nivolumab 480mg q4w up to 1 year.
  Other Names: Ipilimumab 1 mg/kg; Nivolumab 3 mg/kg
  Arms: PHP + IPI1/NIVO3
Drug: IPI3/NIVO1 — Patients will be treated with 4 cycles of intravenous (i.v.) infusion with ipilimumab 3mg/kg and nivolumab 1mg/kg q3w followed by continued i.v. nivolumab 480mg q4w up to 1 year.
  Other Names: Ipilimumab 3 mg/kg; Nivolumab 1 mg/kg
  Arms: IPI3/NIVO1

SUMMARY:
Uveal melanoma is the most common primary intraocular malignancy in adults. Despite successful control of the primary tumor, metastatic disease will develop in approximately 35%-50% of the patients within 10 years. The liver is the most common site for metastases, and about 50% of the patients will have isolated liver metastases. These metastases are generally refractory to systemic chemotherapy and the median survival for patients with liver metastases is about 6 months. Regardless of treatment, the mortality rate is approximately 90% at 2 years with only about 1% of the patients surviving more than 5 years.

The primary objective with this study is to evaluate progression-free survival in patients with uveal melanoma liver metastases randomized to either percutaneous hepatic perfusion (PHP) in combination with ipilimumab and nivolumab or ipilimumab and nivolumab only. Secondary objectives include further efficacy and safety analysis, as well as biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years.
2. Signed informed consent.
3. ECOG performance status of 0 or 1.
4. Histologically or cytologically confirmed liver metastasis of uveal melanoma.
5. Measurable disease by computed tomography (CT) per RECIST 1.1 criteria with at least one target lesion identified in the liver.
6. No previous treatment for uveal melanoma metastases, except patients that have confirmed progression on tebentafusp, or after surgical resection or ablative treatments (e.g., radiofrequency ablation or stereotactic body radiation therapy).
7. Patient deemed suitable for percutaneous hepatic perfusion.
8. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female patients of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Life expectancy of less than 6 months.
2. More than 50% of the liver volume replaced by tumor as measured by CT.
3. Extrahepatic disease as measured by CT of thorax and abdomen.
4. History of congestive heart failure, active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), significant arrhythmias and severe valvular disease that precludes the use of general anesthesia.
5. History or evidence of clinically significant pulmonary disease e.g. severe COPD that precludes the use of general anesthesia.
6. Patients who are unable to undergo general anesthesia for any reason.
7. Reduced renal function defined as S-Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockroft and Gault formula.
8. Reduced hepatic function (defined as AST, ALT, bilirubin>2.5*ULN and PK-INR>1.5) or medical history of liver cirrhosis (Child-Pugh Class B or C) or evidence of portal hypertension by history, endoscopy or radiology.
9. Hemoglobin <90 g/L or platelets <100x109/L or neutrophils <1.5x109/L.
10. Use of live vaccines four weeks before or after the last study treatment.
11. History of severe reactions to monoclonal antibodies, melphalan, heparin or iodine contrast.
12. Known human immunodeficiency virus (HIV) infection, acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C.
13. Active autoimmune disease or a documented history of autoimmune disease requiring systemic immunomodulatory treatment. Diabetes, rheumatoid arthritis, psoriasis, atopic dermatitis and hypothyroidism are excepted.
14. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
15. Concomitant therapy with any other anti-cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs.
16. Has a known additional malignancy that is progressing or requires active treatment.
17. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of study drug.
18. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 24 month
  The primary objective is to evaluate progression-free survival in patients with uveal melanoma hepatic dominant metastases randomized to either percutaneous hepatic perfusion (PHP) in combination with IPI1/NIVO3 or the combination of IPI3/NIVO1 only

SECONDARY OUTCOMES:
Adverse events | 24 month
  Frequency and severity of AEs and SAEs graded according to the NCI CTCAE v5.0.
Overall response rate | 24 month
  Evaluation of objective response rate (ORR), defined as the percentage of patients achieving a confirmed complete or partial response, as defined by RECIST version 1.1 criteria
Clinical benefit rate | 24 month
  Evaluation of clinical benefit rate (CBR), defined as the percentage of patients achieving confirmed SD or any confirmed CR or PR. As defined by RECIST version 1.1 criteria
Hepatic progression-free survival | 24 month
  Evaluation of hepatic PFS (hPFS), defined as the time-to-event defined by the first documented disease progression in the liver or death due to any cause, whichever occurs first, from randomization. hPFS will be determined based on tumor assessment using RECIST version 1.1 criteria.
Overall survival | 24 month
  Evaluation of overall survival (OS), defined as the time from randomization to death from any cause.
Melanoma-specific survival | 24 month
  Evaluation of melanoma-specific survival (MSS), defined as the time from randomization to death from uveal melanoma
Duration of response | 24 month
  Evaluation of duration of response (DOR), defined as the time to first documented progression or death due to underlying cancer from the first document CR or PR
Quality of Life as assessed by FACT-G | 24 month
  Evaluation of QoL using The Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire, where overall scores for FACT-G and the sub scales physical (PWB), social (SWB), emotional (EWB), and functional well-being (FWB) will be reported.
Quality of Life as assessed by EQ-5D-5L | 24 month
  Evaluation of QoL using EQ-5D-5L where EQ-VAS (0-100) will be reported

OTHER OUTCOMES:
ctDNA zero-conversion rate at 24 weeks | 24 weeks
  ctDNA zero-conversion rate at 24 weeks, defined as the percentage of patients that at 24 weeks have no measurable ctDNA levels compared to baseline sample
Biomarker discovery | 24 month
  Predictive and prognostic biomarker discovery

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, Professor, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Karolinska University Hospital,, Stockholm
  - Norrland University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No